CLINICAL TRIAL: NCT01876810
Title: Testing the PPAR Hypothesis of Nicotine Dependence in Humans: Gemfibrozil as a Novel Treatment for Tobacco Addiction
Brief Title: Initial Screening of Gemfibrozil as a Novel Treatment for Tobacco Addiction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 082/2012; NCT01900145 (obsolete NCT alias)
Record Dates: First submitted 2013-06-06; First posted 2013-06-13 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Nicotine Dependence
Keywords: Gemfibrozil; Nicotine Dependence; Smoking; Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Gemfibrozil; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemfibrozil (Experimental): 600 mg of gemfibrozil (one capsule) twice daily for two weeks.
  Interventions: Drug: Gemfibrozil
- Placebo pill (Placebo Comparator): One lactose pill twice a day for two weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemfibrozil — 600 mg of gemfibrozil (one capsule) twice daily for two weeks.
  Other Names: Lopid
  Arms: Gemfibrozil
Drug: Placebo — One lactose pill twice a day for two weeks.
  Other Names: Lactose
  Arms: Placebo pill

SUMMARY:
The purpose of this study is to investigate the effect of gemfibrozil on nicotine reinforcement and cue-elicited craving. Other objectives of this study include screening for the ability of gemfibrozil to aid smoking abstinence during a brief quit attempt and examining the validity of using laboratory measures of tobacco dependence to predict smoking abstinence. It is hypothesized that gemfibrozil will result in diminished nicotine reinforcement, an attenuated response to smoking cues, and an increase in smoking abstinence compared with placebo. It is also hypothesized that the laboratory measures will prove valid in predicting abstinence.

DETAILED DESCRIPTION:
Animal studies have shown that drugs acting as agonists at alpha-type peroxisome proliferator-activated receptors (PPARα) suppress nicotine self-administration, attenuate relapse to nicotine-seeking behavior in the reinstatement model, and block nicotine-induced neuronal firing and dopamine release in reward pathways of the brain. These results have been demonstrated with synthetic PPARα agonists and with fibrate drugs (clofibrate, fenofibrate), which are used clinically to treat elevated cholesterol and triglycerides levels. Thus, PPARα is a potential target for the treatment of tobacco addiction. This is the first human study to investigate whether a fibrate drug (gemfibrozil, Lopid®) can reduce nicotine reward and aid smokers in becoming tobacco abstinent.

The objectives of this study are:

1. to investigate the effect of gemfibrozil on laboratory measures of nicotine reinforcement and cue-elicited craving
2. to screen for the ability of gemfibrozil to aid smoking abstinence during a brief quit attempt
3. to examine the validity of using laboratory measures of tobacco dependence to predict smoking abstinence and possible gemfibrozil-related increases in smoking abstinence

This outpatient study will be conducted at the Center for Addiction and Mental Health (CAMH) in Toronto, Canada. This site will enroll 40 adult smokers who intend to quit smoking in the next 3 months.

The study is a double-blind, placebo-controlled, crossover design comparing the effects of gemfibrozil and placebo. The study will comprise two 2-week medication phases with a washout period of at least one week. At the end of the first medication week laboratory measures will be taken and during the second medication week participants will make a quit attempt and abstinence will be assessed.

Outcome measures include laboratory assessments of nicotine reinforcement and smoking cue reactivity. The measure of nicotine reinforcement is the percentage of nicotine cigarette puffs chosen during a forced-choice task. Measures of cue reactivity include tobacco craving, mood, and autonomic responsivity. Other measures are days of smoking abstinence during the quit-attempt weeks. Abstinence is assessed by self-reports of no smoking and by breath carbon monoxide < 5 ppm on clinic visits. Other assessments of abstinence include self-reported tobacco craving and withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* 19-65 year old males and females
* smoking at least 10 cigarettes per day for at least 2 years
* intend to quit smoking within the next 3 months
* medically and psychologically healthy as determined by screening criteria

Exclusion Criteria:

* currently attempting to quit smoking
* treatment for tobacco addiction in the past 3 months
* use of nicotine replacement products, bupropion, or varenicline in the past 3 months as an aid to quit or reduce smoking
* use of any oral tobacco product in the past 3 months
* history of drug or alcohol dependence within last 5 years
* consumption of more than 15 alcoholic drinks per week on average during the past month
* use of any illicit drug more than once per week on average during the past month
* current use of gemfibrozil or other fibrate medication
* current use of any medication that is contraindicated for gemfibrozil or that would interfere with the protocol in the opinion of MAI/QI. This includes, but is not limited to, anticoagulants, statins, other fibrates, other lipid-lowering agents such as niacin or herbal remedies, and any oral or injected medications for diabetes.
* any pre-existing gall-bladder disease or operation in the past 12 months
* any history of or current cardiovascular, liver, hepatic or renal disease
* diabetes
* pregnant, nursing, or become pregnant during the study
* use of psychoactive drugs or medications as revealed by urine toxicology

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Centre of Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was excluded after enrollment after disclosure of a mental illness which is an exclusion criteria.
Groups:
- Gemfibrozil/Placebo: Participants received 600 mg of gemfibrozil (one capsule) twice daily for two weeks. Then a washout period of 1 week of no medication. Then they received 1 capsule of placebo twice daily for 2 weeks
- Placebo/Gemfibrozil: Participants received 1 capsule of placebo for 2 weeks. Then a washout period of 1 week of no medication. Then they received 600 mg of gemfibrozil (one capsule) twice daily for two weeks.
Period: Overall Study
Arm/Group | Gemfibrozil/Placebo | Placebo/Gemfibrozil
Started | 14 | 14
Completed | 14 | 13
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 600 mg of gemfibrozil (one capsule) twice daily for two weeks.
  Gemfibrozil: 600 mg of gemfibrozil (one capsule) twice daily for two weeks. or One lactose pill twice a day for two weeks.
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Self-report of No Smoking and Breath Carbon Monoxide of <5 PPM During Quit-attempt Weeks
Description: the number of days of no smoking was calculated for each participant. Abstinence was verified by daily Self-reports of no smoking and breath carbon monoxide < 5 ppm
Time Frame: 1 week in each phase
Measure: Mean (Standard Error); unit: days
Groups:
- Gemfibrozil: Participants taking Gemfibrozil: 600 mg of gemfibrozil (one capsule) twice daily for two weeks during the 1st phase of the study or during the second phase after a washout period .
- Placebo: Participants taking Placebo (one capsule) twice daily for two weeks during the 1st phase of the study or during the second phase after a washout period.
Arm/Group | Gemfibrozil | Placebo
Number analyzed (Participants) | 27 | 27
days | 0.2 (0.1) | 0 (0)
Statistical Analysis 1: Comparison: Gemfibrozil; Test type: Superiority or Other; p = 0.1, t-test, 2 sided — For all analyses, results are considered significant at p<.05; Mean Difference (Final Values) = 0.2, Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.1, t-test, 2 sided — For all analyses, results were considered significant at p< 0.05; Median Difference (Final Values) = 0.0, Standard Error of Mean 0.0

2. Secondary Outcome: The Percentage of Choice of Nicotinized Cigarettes After 1 Week of Treatment
Description: Percentage of choice of Nicotinized cigarettes was calculated for each participant during the lab session which took place after 1 week of treatment.
  Each session started with participants taking four puffs of their preferred-brand cigarette to standardize the time from last nicotine exposure. Participants were asked to complete some questionnaires at baseline. Then, they were asked to relax for 30 min listening to music or reading. Four exposure trials followed that were separated by 30 min of relaxation. In each exposure trial, participants took four puffs of a Nicotinized (A) or Denicotinized (less than 0.05 mg nicotine.) (B) cigarette in the order of ABAB or BABA. Cigarettes were color-coded. Participants then began four choice trials separated by 30 min of relaxation. In each trial, participants chose any combination of 4 puffs from the two cigarettes.
Time Frame: during the lab forced choice paradigm after 1 week of treatment
Measure: Mean (Standard Error); unit: percentage of choice of nicotinized ciga
Groups:
- Gemfibrozil: Participants taking Gemfibrozil: 600 mg of gemfibrozil (one capsule) twice daily for two weeks during the 1st phase of the study or during the second phase after the washout period.
- Placebo Group: Participants taking Placebo (one capsule) twice daily for two weeks during the 1st phase of the study or during the second phase after the washout period.
Arm/Group | Gemfibrozil | Placebo Group
Number analyzed (Participants) | 27 | 27
percentage of choice of nicotinized ciga | 0.775 (0.034) | 0.77 (0.05)
Statistical Analysis 1: Comparison: Gemfibrozil; Test type: Superiority or Other; p = 0.9, t-test, 2 sided — For all analyses, results were considered significant at p< 0.05; Mean Difference (Final Values) = 0.77, Standard Error of Mean 0.034
Statistical Analysis 2: Comparison: Placebo Group; Test type: Superiority or Other; p = 0.9, t-test, 2 sided — For all analyses, results were considered significant at p< 0.05; Mean Difference (Final Values) = 0.77, Standard Error of Mean 0.05

3. Other Pre Specified Outcome: Cue- Reactivity Visual Analogue Scale for Craving After 1 Week of Treatment
Description: In this study, each session started with participants taking four puffs of their preferred-brand cigarette to standardize the time from last nicotine exposure. Participants were then seated in a comfortable chair and completed the baseline Visual Analogue Scale for craving 0-100 mm (The higher the number the more is the craving). The smoking cue was a pack of cigarettes and a lighter. Participants were instructed to light the cigarette without puffing and hold it for 30 sec while the physiological recordings were measured. Then the participant was asked to extinguish the cigarette. The neutral cue was an unsharpened pencil, a notepad, and a sharpener. Participants were instructed to sharpen the pencil and hold it as if writing for 30 sec. Participants completed the Visual Analogue Scale for craving during the cue, and 15 and 30 min after cue presentation.
Time Frame: during the lab Cue- reactivity paradigm after 1 week of treatment
Population: participants self-reportd Visual analogue scale (0-100 mm) for craving at the time of presenting the smoking cue. The higher the number on the scale, the more is the craving
Measure: Mean (Standard Error); unit: units on a scale: from 0-100 mm
Groups:
- Gemfibrozil: Participants taking Gemfibrozil 600 mg (one capsule twice daily) for two weeks during the 1st phase of the study or during the second phase after the washout period.
Arm/Group | Gemfibrozil | Placebo Group
Number analyzed (Participants) | 27 | 27
units on a scale: from 0-100 mm | 51 (32.7) | 44 (27.4)
Statistical Analysis 1: Comparison: Gemfibrozil; Test type: Superiority or Other; p = 0.4, ANOVA; Repeated-measures ANOVA on Drug X Cue X Time were used; Mean Difference (Final Values) = 51.3, Standard Error of Mean 31.7 — participants self-reportd VAS craving at the time of neutral cue presentation
Statistical Analysis 2: Comparison: Placebo Group; Test type: Superiority or Other; p = 0.4, ANOVA — For all analyses, results were considered significant at p< 0.05; Repeated-measures ANOVA on Drug X Cue X Time were used; Mean Difference (Final Values) = 43.7, Standard Error of Mean 26.5

ADVERSE EVENTS:
Time Frame: The side effects were collected for each participant over six weeks from the start of treatment (2 weeks gemfibrozil/or placebo), 1 week washout period, (2 weeks gemfibrozil/or placebo), and 1 week after completion of the study.
Groups:
- Gemfibrozil/Placebo: 600 mg of gemfibrozil (one capsule) twice daily for two weeks.
  Participants taking Gemfibrozil: 600 mg of gemfibrozil (one capsule) twice daily for two weeks during the 1st phase of the study followed by a the washout period. Then they received 1 capsule of placebo twice daily for 2 weeks
- Placebo/Gemfibrozil: One lactose pill twice a day for two weeks.
  Participants taking Placebo (one capsule) twice daily for two weeks during the 1st phase of the study followed by a the washout period. Then they received 1 capsule of gemfibrozil twice daily for 2 weeks
Arm/Group | Gemfibrozil/Placebo | Placebo/Gemfibrozil
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 8/14 | 6/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemfibrozil/Placebo (N=14) | Placebo/Gemfibrozil (N=13)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Change in appetite (Gastrointestinal disorders) | 2 (2) | 4 (4)
stomach upset (Gastrointestinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes